CLINICAL TRIAL: NCT05112393
Title: Development and Validation of Creatinine-Based Estimates of the Glomerular Filtration Rate Equation From Chromium EDTA Imaging in the Multi-racial Malaysian Population
Brief Title: Development and Validation of Creatinine-Based Estimates of the Glomerular Filtration Rate Equation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: eGFR MY
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Renal Function Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development Cohort: Half of the data will be randomized into development cohort by using a random number generated in Microsoft Excel. This cohort aim to develop a new estimating Glomerular Filtration Rate (eGFR) equation that produce accurate eGFR specifically in Malaysian multiracial population.
  Interventions: Other: Development of new estimating Glomerular Filtration Rate (eGFR) equation
- Validation Cohort: Half of the data will be randomized into development cohort by using a random number generated in Microsoft Excel. This cohort aim to validate the newly developed estimating Glomerular Filtration Rate (eGFR) equation.
  Interventions: Other: Validation of new estimating Glomerular Filtration Rate (eGFR) equation

INTERVENTIONS:
Other: Development of new estimating Glomerular Filtration Rate (eGFR) equation — Development Cohort:
  A new estimating Glomerular Filtration Rate(eGFR) equation will be developed by using a nonlinear regression model utilizing a generalized least squares algorithm.
  Groups: Development Cohort
Other: Validation of new estimating Glomerular Filtration Rate (eGFR) equation — Validation Cohort:
  Internal validation will be performed by comparing bias, precision and accuracy of the new equations and the other established equations to the measured GFR.
  Groups: Validation Cohort

SUMMARY:
This study aim to recruit all Electronic Medical Record of patients who underwent for 51chromium ethylenediamine tetra acetic acid (51Cr-EDTA) imaging at the Nuclear Medicine Centre, University Malaya Medical Centre from September 2016 to September 2021. The data that collected will be analyzed to develop and validate a new equation to estimate Glomerular Filtration Rate that specifically for Malaysian multiracial population.

DETAILED DESCRIPTION:
List of patients who underwent for 51Cr EDTA imaging at the Nuclear Medicine Centre, University Malaya Medical Centre from September 2016 to September 2021 will be obtained from relevant department. All patient's Electronic Medical Record (EMR) will be evaluated for recruitment into the study.

Demographics data of the patients that will be collected include age, gender, height, weight, and ethnicity. The clinical data that will be collected include CKD aetiology, background comorbidities, and vitals sign and laboratory data includes the renal function test. The 51Cr- EDTA readings were also recorded.

If there are multiple measurements of scans performed, the latest 51Cr-EDTA taken. The renal function test must be within three months of when the 51Cr-EDTA imaging was conducted.

Patients will be randomized into a development and validation cohort using a random number generated in Microsoft Excel. In the development cohort, a new equation will be developed using a nonlinear regression model utilizing a generalized least squares algorithm. Internal validation will be performed in the validation cohort, by comparing the bias, precision, and accuracy of the new equations and the other established equations to the measured GFR.

ELIGIBILITY:
Inclusion Criteria:

* Electronic Medical Records of patient scheduled for 51Cr EDTA imaging at the Nuclear Medicine Centre, University Malaya Medical Centre from September 2016 to September 2021
* Age 16-year-old and above

Exclusion Criteria:

* Electronic Medical Records of patients with missing data.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Electronic Medical Records of patient scheduled for 51Cr EDTA imaging at the Nuclear Medicine Centre, University Malaya Medical Centre from September 2016 to September 2021
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
New equation to estimate GFR that can be used specifically in Malaysian multiracial population | From 1st December 2021 to 31st December 2022
  New equation that has its own ethnic coefficient that can produce accurate result in Malaysia multiracial population

CONTACTS AND LOCATIONS:
Overall Officials: Ina Ismiarti Shariffuddin, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Diego E, Castro P, Soy D, Poch E, Nicolas JM. Predictive performance of glomerular filtration rate estimation equations based on cystatin C versus serum creatinine values in critically ill patients. Am J Health Syst Pharm. 2016 Feb 15;73(4):206-15. doi: 10.2146/ajhp140852. PMID 26843497
- [Background] Bragadottir G, Redfors B, Ricksten SE. Assessing glomerular filtration rate (GFR) in critically ill patients with acute kidney injury--true GFR versus urinary creatinine clearance and estimating equations. Crit Care. 2013 Jun 15;17(3):R108. doi: 10.1186/cc12777. PMID 23767877
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Rule AD, Teo BW. GFR estimation in Japan and China: what accounts for the difference? Am J Kidney Dis. 2009 Jun;53(6):932-5. doi: 10.1053/j.ajkd.2009.02.011. No abstract available. PMID 19463761
- [Background] Matsuo S, Yasuda Y, Imai E, Horio M. Current status of estimated glomerular filtration rate (eGFR) equations for Asians and an approach to create a common eGFR equation. Nephrology (Carlton). 2010 Jun;15 Suppl 2:45-8. doi: 10.1111/j.1440-1797.2010.01313.x. PMID 20586948
- [Background] Zelnick LR, Leca N, Young B, Bansal N. Association of the Estimated Glomerular Filtration Rate With vs Without a Coefficient for Race With Time to Eligibility for Kidney Transplant. JAMA Netw Open. 2021 Jan 4;4(1):e2034004. doi: 10.1001/jamanetworkopen.2020.34004. PMID 33443583
- [Background] Matsuo S, Imai E, Horio M, Yasuda Y, Tomita K, Nitta K, Yamagata K, Tomino Y, Yokoyama H, Hishida A; Collaborators developing the Japanese equation for estimated GFR. Revised equations for estimated GFR from serum creatinine in Japan. Am J Kidney Dis. 2009 Jun;53(6):982-92. doi: 10.1053/j.ajkd.2008.12.034. Epub 2009 Apr 1. PMID 19339088
- [Background] Jeong TD, Lee W, Yun YM, Chun S, Song J, Min WK. Development and validation of the Korean version of CKD-EPI equation to estimate glomerular filtration rate. Clin Biochem. 2016 Jun;49(9):713-719. doi: 10.1016/j.clinbiochem.2016.01.023. Epub 2016 Mar 9. PMID 26968101
- [Background] Praditpornsilpa K, Townamchai N, Chaiwatanarat T, Tiranathanagul K, Katawatin P, Susantitaphong P, Trakarnvanich T, Kanjanabuch T, Avihingsanon Y, Tungsanga K, Eiam-Ong S. The need for robust validation for MDRD-based glomerular filtration rate estimation in various CKD populations. Nephrol Dial Transplant. 2011 Sep;26(9):2780-5. doi: 10.1093/ndt/gfq815. Epub 2011 Feb 28. PMID 21357214
- [Background] Assadi M, Eftekhari M, Hozhabrosadati M, Saghari M, Ebrahimi A, Nabipour I, Abbasi MZ, Moshtaghi D, Abbaszadeh M, Assadi S. Comparison of methods for determination of glomerular filtration rate: low and high-dose Tc-99m-DTPA renography, predicted creatinine clearance method, and plasma sample method. Int Urol Nephrol. 2008;40(4):1059-65. doi: 10.1007/s11255-008-9446-4. Epub 2008 Aug 9. PMID 18690545
- [Background] Liu X, Qiu X, Shi C, Huang H, Huang J, Li M, Lou T. Modified glomerular filtration rate-estimating equations developed in asiatic population for chinese patients with type 2 diabetes. Int J Endocrinol. 2014;2014:521071. doi: 10.1155/2014/521071. Epub 2014 Mar 5. PMID 24734043
- [Background] Liao Y, Liao W, Liu J, Xu G, Zeng R. Assessment of the CKD-EPI equation to estimate glomerular filtration rate in adults from a Chinese CKD population. J Int Med Res. 2011;39(6):2273-80. doi: 10.1177/147323001103900624. PMID 22289543
- [Background] Ma YC, Zuo L, Zhang CL, Wang M, Wang RF, Wang HY. Comparison of 99mTc-DTPA renal dynamic imaging with modified MDRD equation for glomerular filtration rate estimation in Chinese patients in different stages of chronic kidney disease. Nephrol Dial Transplant. 2007 Feb;22(2):417-23. doi: 10.1093/ndt/gfl603. Epub 2006 Oct 19. PMID 17053082
- [Background] Madala ND, Nkwanyana N, Dubula T, Naiker IP. Predictive performance of eGFR equations in South Africans of African and Indian ancestry compared with (9)(9)mTc-DTPA imaging. Int Urol Nephrol. 2012 Jun;44(3):847-55. doi: 10.1007/s11255-011-9928-7. Epub 2011 Mar 5. PMID 21373844
- [Background] Jalalonmuhali M, Kok Peng N, Soo Kun L. Comparative Performance of Creatinine-Based Estimated Glomerular Filtration Rate Equations in the Malays: A Pilot Study in Tertiary Hospital in Malaysia. Int J Nephrol. 2017;2017:2901581. doi: 10.1155/2017/2901581. Epub 2017 Jun 18. PMID 28702264
- [Background] Jalalonmuhali M, Lim SK, Md Shah MN, Ng KP. MDRD vs. CKD-EPI in comparison to 51Chromium EDTA: a cross sectional study of Malaysian CKD cohort. BMC Nephrol. 2017 Dec 13;18(1):363. doi: 10.1186/s12882-017-0776-2. PMID 29237422
- [Background] Jalalonmuhali M, Elagel SMA, Tan MP, Lim SK, Ng KP. Estimating Renal Function in the Elderly Malaysian Patients Attending Medical Outpatient Clinic: A Comparison between Creatinine Based and Cystatin-C Based Equations. Int J Nephrol. 2018 May 13;2018:3081518. doi: 10.1155/2018/3081518. eCollection 2018. PMID 29862077
- [Background] Md Ralib A, Mohd Hanafiah FN, Abd Rashid I, Abd Rahim MS, Dzaharudin F, Mat Nor MB. Development and Validation of Creatinine-Based Estimates of the Glomerular Filtration Rate Equation from 99mTc-DTPA Imaging in the Malaysian Setting. Int J Nephrol. 2021 Sep 8;2021:3465472. doi: 10.1155/2021/3465472. eCollection 2021. PMID 34540290